CLINICAL TRIAL: NCT07405996
Title: Referral of Patients With Biological Abnormalities to an Emergency Department : ORA
Brief Title: Referral of Patients With Biological Abnormalities to an Emergency Department
Acronym: ORA
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-06-Obs-CHRMT
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Biological Abnormality; Emergency Department Visit; General Practitioner

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Biological testing is an essential part of general medical practice and plays a role in 60% to 70% of diagnoses. 68.5% of prescriptions are written by general practitioners, and one in seven general medical consultations ends with a prescription for biological testing. The study of patient trajectories is a recent emerging topic in the literature, encompassing general concepts. The angle most often taken is medico-economic and focused on specific chronic conditions such as diabetes, cancer, or cardiovascular disease. To our knowledge, there are a number of referrals to emergency departments by general practitioners for patients with biological abnormalities. However, to our knowledge, no study to date has attempted to quantify these specific referrals.

DETAILED DESCRIPTION:
want to establish a register of biological anomaly referrals by general practitioners to emergency departments. This study will enable us to estimate the number of patients whose referral could have been handled differently, allowing us to develop dedicated care pathways, specialized training in outpatient settings, or targeted communications, ultimately leading to better patient referral and reducing inappropriate use of emergency services.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting at an emergency department participating in the IOA (nurse coordinating reception) system with the reason for referral "Abnormal laboratory results.

Exclusion Criteria:

* minor patients (<18 years old)
* expression of the patient's opposition to the collection of data relating to their hospital stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient presenting at an emergency department participating in the IOA (nurse coordinating reception) system with the reason for referral "Abnormal laboratory results.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Type of biological abnormality and severity level | Immediately upon admission to the emergency room
  The primary evaluation criterion is the type of biological abnormality sent to the emergency department and its severity (depth or elevation).

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz-Thionville, Metz, France, France

IPD SHARING:
Plan to Share IPD: No